CLINICAL TRIAL: NCT05702268
Title: A Randomized, Double-blind, Placebo-controlled Phase II Trial Evaluating the Safety, Efficacy, Pharmacokinetics, and Pharmacodynamics of ICP-332 in Moderate-to-severe Atopic Dermatitis
Brief Title: Pharmacodynamic Blood Characteristics of ICP-332 in Patients With Moderate to Severe Atopic Dermatitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICP-CL-00602
Record Dates: First submitted 2023-01-10; First posted 2023-01-27 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Moderate to Severe Atopic Dermatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-dose (Experimental): 40 mg ICP-332 tablet 3 tablets, once a day
  Interventions: Drug: ICP-332
- Low-dose (Experimental): 40 mg ICP-332 2 tablets + 1 placebo tablet once daily
  Interventions: Drug: ICP-332; Drug: ICP-332 Placebo
- Blank control (Placebo Comparator): Placebo 3 tablets once daily
  Interventions: Drug: ICP-332 Placebo

INTERVENTIONS:
Drug: ICP-332 — Tablet, 40 mg
  Arms: High-dose; Low-dose
Drug: ICP-332 Placebo — Tablets, in appearance, size, color, dosage form, packaging, instructions, labels and other aspects of the corresponding specifications of ICP-332.
  Arms: Blank control; Low-dose

SUMMARY:
The investigator, the subject, and the sponsor's project team will remain blind throughout the study. Subjects will be randomly assigned to one of the three treatment groups at a ratio of 1:1:1 to be given the drug once a day for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥18 years and ≤75 years.
2. A clinical diagnosis of atopic dermatitis or eczema was made at least 1 year prior to D1, and atopic dermatitis was identified at screening visit (according to Williams criteria).
3. During screening and baseline, were defined as meeting the moderate and severe AD criteria as assessed by the researchers.
4. Documented history of inadequate response to topical corticosteroids (TCS) or topical calcineurin inhibitors (TCI) , or other medically unrecommended topical therapy.
5. Able and willing to use an additive free mild emollient twice a day for at least 7 days prior to baseline and for the duration of the study.
6. The serum pregnancy test of all female subjects at screening visit was negative, and the urine pregnancy test of all fertile female subjects at baseline visit was negative before first dosing.
7. Subjects must voluntarily sign and date informed consent prior to the commencement of any screening or study specific procedures.
8. Subject is willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.
9. Fertile women (WOCBP) menstruation must occur during the screening period and consent to use a supplementary screen contraceptive method in combination with a highly effective contraceptive method during the study period and for 90 days after the last use of the study drug .Male subjects must be willing not to donate sperm during this period.

Exclusion Criteria:

1. Pregnant female subjects and nursing female subjects.
2. Subjects who had an active skin disease or skin infection that required systemic treatment or would interfere with the proper assessment of AD.
3. Current or previous infection history, including a history of herpes; Known history of invasive infection; Chronic recurrent infection and/or active invasive infection. Known immunodeficiency syndrome; Subjects with tuberculosis; Non skin related active infection.
4. Active HBV, HCV or HIV, syphilis infection.
5. Potential medical diseases or problems, including but not limited to the following: clinically relevant or significant ECG abnormalities; History of moderate to severe congestive heart failure, recent cerebrovascular accident, myocardial infarction or coronary stent implantation, or uncontrolled hypertension; Have received organ transplantation; A history of gastrointestinal perforation, diverticulitis, or a significant increased risk of gastrointestinal perforation according to the investigator's judgment; Diseases that may interfere with drug absorption; Subjects suffering from any malignant tumor before screening.
6. Except for atopic dermatitis, he has any clinically significant disease history or other clinically significant systemic diseases.
7. Received the specified treatment plan within the specified time frame.
8. The time from the last use of powerful CYP3A inhibitor or inducer to the first trial medication is less than 5 clearance half-life, or it is planned to take powerful CYP3A inhibitor or inducer at the same time during this study.
9. Those with a history of drug or alcohol abuse in the 6 months prior to baseline visit (as determined by the investigator).
10. During the screening period before the first administration of the study drug (baseline visit), the abnormal laboratory values met at least one of the specified standards.
11. The investigator considers for any reason that the subject is not suitable for participation in the study to receive ICP-332.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-03-18 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | Up to 24 weeks
Systolic and Diastolic Blood Pressure | Up to 24 weeks
Pulse Rate | Up to 24 weeks
Electrocardiogram (ECG) QT Interval | Up to 24 weeks
Number of participants with treatmentrelated adverse events as assessed by CTCAE v4.0 | Up to 24 weeks

SECONDARY OUTCOMES:
Percentage change of EASI score from baseline in week 4 | 4 weeks

CONTACTS AND LOCATIONS:
Locations (28):
- China (28):
  - Beijing Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Second Hospital of the Army Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The Affiliated Hospital of Chengde Medical College, Chengde, Hebei
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Nanyang First People's Hospital, Nanyang, Henan
  - Shiyan City People's Hospital, Shiyan, Hubei
  - Wuhan University People's Hospital, Wuhan, Hubei
  - Changzhou First People's Hospital, Changzhou, Jiangsu
  - Wuxi Second People's Hospital, Wuxi, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Dermatology Hospital, Shanghai, Shanghai Municipality
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - The Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Suining Central Hospital, Suining, Sichuan
  - Affiliated Hospital of Tianjin Academy of Traditional Chinese Medicine, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Hangzhou Third People's Hospital, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Jiaxing First Hospital, Jiaxing, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

REFERENCES:
- [Derived] Xu J, Zhang L, Liang Y, Ji C, Xu A, Li Z, Li L, Lei T, Zhang C, Chen R, Tao X, Zhang R, Fang H, Zheng J, Yang W, Zhang G, Duan X, Ding Y, Yin W, Zhou W, Fan D, Du Y. Safety and Efficacy of ICP-332 for Moderate to Severe Atopic Dermatitis: A Phase 2 Randomized Clinical Trial. JAMA Dermatol. 2026 Jan 14. doi: 10.1001/jamadermatol.2025.5295. Online ahead of print. PMID 41533373